CLINICAL TRIAL: NCT03633786
Title: Evaluation of Robot-assisted Versus Standard Laparoscopic Approach for the Surgical Treatment of Deep Infiltrating Endometriosis
Brief Title: Robot-assisted Versus Standard Laparoscopic Approach for the Surgical Treatment of Deep Infiltrating Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Renato Seracchioli, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VINCENDO-01
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Endometriosis
Keywords: endometriosis; robot-assisted surgery; standard laparoscopic surgery
MeSH Terms: conditions — Endometriosis | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: standard laparoscopic surgery (Other): patients affected by deep infiltrating endometriosis undergoing standard laparoscopic surgery; assessment of sexual function; assessment of bowel symptoms; assessment of urinary symptoms
  Interventions: Procedure: standard laparoscopic surgery; Diagnostic Test: assessment of sexual function; Diagnostic Test: assessment of bowel symptoms; Diagnostic Test: assessment of urinary symptoms
- Group B: robot-assisted surgery (Other): patients affected by deep infiltrating endometriosis undergoing robot-assisted surgery; assessment of sexual function; assessment of bowel symptoms; assessment of urinary symptoms
  Interventions: Procedure: robot-assisted surgery; Diagnostic Test: assessment of sexual function; Diagnostic Test: assessment of bowel symptoms; Diagnostic Test: assessment of urinary symptoms

INTERVENTIONS:
Procedure: standard laparoscopic surgery — removal of endometriotic lesions with laparoscopic instruments (KARL STORZ Gesellschaft mit beschränkter Haftung & Co., Tuttlingen, Germany) using 4 transperitoneal abdominal accesses and trocars from 5 to 12 mm
  Arms: Group A: standard laparoscopic surgery
Procedure: robot-assisted surgery — removal of endometriotic lesions with da Vinci Xi robotic system (Intuitive Surgical Inc., Sunnyvale, CA, USA), using 5 transperitoneal abdominal accesses and trocars from 8 and 12 mm.
  The robotic mechanical arms are associated with the 8 mm abdominal trocars to allow intervention by the first operator, with the aid of a surgical console.
  Arms: Group B: robot-assisted surgery
Diagnostic Test: assessment of sexual function — assessment of sexual function using a validate questionnaire (Female Sexual Function Index (FSFI)), before and 3 months after surgery
Diagnostic Test: assessment of bowel symptoms — assessment of bowel symptoms using a validated questionnaire (Knowles-Eccersley-Scott-Symptom Questionnaire (KESS)), before and 3 months after surgery
Diagnostic Test: assessment of urinary symptoms — assessment of urinary symptoms using a validated questionnaire (Bristol Female Lower Urinary Tract Symptoms (BFLUTS)), before and 3 months after surgery

SUMMARY:
Deep infiltrating endometriosis (DIE) is a severe form of endometriosis in which lesions affect retroperitoneal tissue and pelvic organs wall. It is often a cause of significant pain (dysmenorrhea, dysuria, dyspnea, dyspareunia and chronic pelvic pain) and infertility, drastically reducing patients' quality of life.

Surgical therapy with complete removal of endometriotic lesions is often necessary when the disease is resistant to medical therapy.

The minimally invasive surgical approach has proved to be the most advantageous.

Over time, there has been a growing use in the gynecological field of robot-assisted laparoscopic surgery.

Several clinical cases and retrospective studies on robotic surgery for DIE have highlighted favorable surgical outcomes, with the exception of operative times, compared to standard laparoscopic approach.

However, a randomized control studies comparing surgical outcomes and postoperative pelvic organs function in women with DIE submitted to robotic-assisted or conventional laparoscopy is missing.

In order to analyze the real impact of robotic advances the present study sought to assess surgical outcomes and urinary, bowel and sexual functions in women with DIE requiring minimally invasive surgery through robot-assisted or conventional lps approach.

DETAILED DESCRIPTION:
Patients with clinical and trans-vaginal / abdominal ultrasound diagnosis of deep endometriosis, undergoing surgery for the removal of endometriotic lesions are included in the study.

Patients are divided into 2 groups:

Group A: standard laparoscopic approach

Group B: robot-assisted approach

After surgery, patients will be included in the post-operative follow-up, as usual in our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of deep endometriosis based on clinical and transvaginal/transabdominal ultrasound examinations and, when necessary, magnetic resonance
* Patients with indication for removal of endometriosic lesions by standard and robot-assisted laparoscopy
* Obtaining Informed Consent

Exclusion Criteria:

* Contraindications for removal of endometriosic lesions by standard and robot-assisted laparoscopy
* Cardiovascular problems
* Hepatic insufficiency
* Psychiatric diseases
* History of oncologic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative
  Evaluation and comparison of operative time in patients underwent standard laparoscopic or robot-assisted surgery

SECONDARY OUTCOMES:
Length of hospitalization | Up to 4 days: from the date of surgery until the last day of hospitalization
  Evaluation and comparison of the length of hospitalization in patients underwent standard laparoscopic or robot-assisted surgery
Change of haemoglobin levels | 24 hours after surgery
  Evaluation and comparison of the change of haemoglobin levels in patients underwent standard laparoscopic or robot-assisted surgery
Laparotomic conversion rate | Intraoperative
  Evaluation and comparison of laparotomic conversion rate in patients underwent standard laparoscopic or robot-assisted surgery
Evaluation of sexual function | up to three months after surgery
  Evaluation and comparison of sexual function in patients underwent standard laparoscopic or robot-assisted surgery before and after surgery, using the Female Sexual Function Index (FSFI). The FSFI is a validated questionnaire useful to measure sexual functioning in women. It was developed for the specific purpose of assessing domains of sexual functioning (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials. The full scale score range goes from a minimum of 2.0 to a maximum of 36.0.
Evaluation of urinary symptoms | up to three months after surgery
  Evaluation and comparison of urinary symptoms in patients underwent standard laparoscopic or robot-assisted surgery before and after surgery, using the Bristol Female Lower Urinary Tract Symptoms (BFLUTS) questionnaire. It is a validated questionnaire with 3 subscale scores for incontinence symptoms (BFLUTS-IS) (range from 0 to 20), voiding symptoms (BFLUTS-VS) (range from 0 to 12), and filling symptoms (BFLUTS-FS) (range from 0 to 15), with the addition of single subscales for sexual function (BFLUTS-sex) (range from 0 to 6) and quality of life (BFLUTSQoL) (range from 0 to 18).
Evaluation of bowel symptoms | up to three months after surgery
  Evaluation and comparison of bowel symptoms in patients underwent standard laparoscopic or robot-assisted surgery before and after surgery, using the Knowles-Eccersley-Scott-Symptom Questionnaire (KESS). The KESS is a validated questionnaire for diagnosis of constipation. KESS has an added advantage of differentiating between various subtypes of constipation. Total scores can range from 0 (no symptoms) to 39 (high symptom severity). A cut-off score of > 11 indicates constipation.
Evaluation of disease recurrence rate | Up to 12 months after surgery; from date of surgery until the date of first clinical or trans-vaginal/abdominal ultrasound documented recurrence, assessed up to 12 months
  Evaluation and comparison of disease recurrence rate in patients underwent standard laparoscopic or robot-assisted surgery before and after surgery.
  Endometriosis recurrence can have different levels: symptoms recurrence based on patient history (VAS pain score ≥ 5), but no proof of recurrence by imaging and/or surgery; endometriosis recurrence based on non-invasive imaging in patients with or without symptoms; recurrence of histologically proven endometriosis: when the patient is re-operated, endometriosis is visually observed and confirmed histologically.
Complication rate | Intraoperative
  Comparison of standard laparoscopy and robot-assisted surgery concerning intraoperative complication rate in patients affected by deep infiltrating endometriosis
Complication rate | up to three months after surgery; from date of surgery until the date of first documented complication, assessed up to 3 months
  Comparison of standard laparoscopy and robot-assisted surgery concerning complication rate in patients affected by deep infiltrating endometriosis, using Clavien-Dindo Classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, BO, Italy

REFERENCES:
- [Derived] Bafort C, Beebeejaun Y, Tomassetti C, Bosteels J, Duffy JM. Laparoscopic surgery for endometriosis. Cochrane Database Syst Rev. 2020 Oct 23;10(10):CD011031. doi: 10.1002/14651858.CD011031.pub3. PMID 33095458